CLINICAL TRIAL: NCT02172586
Title: A PROBE (Prospective, Randomised, Open-label, Blinded Endpoint) Trial to Investigate the Efficacy and Safety of Telmisartan 40-80 mg Once Daily Compared With Losartan 50-100 mg Once Daily Over a Period of 12 Weeks, and of Telmisartan 80 mg + HCTZ 12.5 mg Once Daily Compared With Losartan 100 mg Once Daily + HCTZ 12.5 mg Once Daily Over a Period of Further 12 Weeks in Mild to Moderate Hypertensive Patients (Grade 1 and Grade 2 WHO-ISH Guidelines 1999)
Brief Title: Telmisartan With or Without Hydrochlorothiazide (HCTZ) Compared With Losartan With or Without HCTZ in Mild to Moderate Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.316
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Losartan; Hydrochlorothiazide

ARMS (4):
- Telmisartan (Experimental)
  Interventions: Drug: Telmisartan
- Telmisartan + Hydrochlorothiazide (Experimental)
  Interventions: Drug: Telmisartan; Drug: Hydrochlorothiazide
- Losartan (Active Comparator)
  Interventions: Drug: Losartan
- Losartan + Hydrochlorothiazide (Active Comparator)
  Interventions: Drug: Losartan; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan; Telmisartan + Hydrochlorothiazide
Drug: Losartan
  Arms: Losartan; Losartan + Hydrochlorothiazide
Drug: Hydrochlorothiazide
  Arms: Losartan + Hydrochlorothiazide; Telmisartan + Hydrochlorothiazide

SUMMARY:
Study to assess the efficacy of telmisartan 40-80 mg once daily compared with losartan 50-100 mg once daily in hypertensive patients evaluated by change from baseline in diastolic blood pressure (DBP) during the last 6 hours of the 24-hour dosing interval, at the end of the 12 weeks period of monotherapy treatment (ABPM - ambulatory blood pressure measurement).

Secondary objectives: Changes from baseline in BP at the end of the monotherapy period of treatment and at the end of the study, evaluated by sphygmomanometric blood pressure measurement and ABPM

Safety:

Incidence of adverse events (AE's); withdrawal due to adverse events; laboratory parameters

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Mild-to-moderate essential hypertension defined as a mean diastolic blood pressure (DBP) ≥ 95 mmHg and < 110 mmHg and systolic blood pressure (SBP) < 180 mmHg measured by manual cuff sphygmomanometer at the end of the wash-out period
* Written informed consent

Exclusion Criteria:

* Nursing, pregnancy or childbearing potential women, post-menopausal women will be enrolled with last menstruation > 1 year prior to start wash-out phase or surgically sterile
* Secondary hypertension
* Malignant hypertension (retinal haemorrhage, exudates or papillary oedema)
* Clinically significant sodium depletion as defined by serum sodium level < 130 mEq/L and/or clinically significant hyperkaliemia as defined by serum potassium level > 5.5 mEq/L or clinically significant hypokaliemia as defined by serum potassium level < 3.0 mEq/L
* Atrial fibrillation or frequent ventricular ectopic beats or other arrhythmias which, in the investigator opinion could compromise patient's participation to the trial
* Congestive heart failure (CHF) (NYHA (New York Heart Association) functional class CHF III-IV)
* Angina pectoris or myocardial infarction
* Cardiac surgery within the past 3 months prior to start the wash-out period
* Stroke within the past 6 months prior to start the wash-out period
* Renal insufficiency defined as creatininaemia > 2mg/dl
* Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post renal transplant, presence of only one functioning kidney
* Liver insufficiency, defined as bilirubinaemia > 2mg/dl and AST (aspartate aminotransferase) or ALT (alanine-aminotransferase) > twice the upper normal range
* Clinically significant metabolic and endocrine disease
* Autoimmune disease
* Previous history of angioedema
* Body mass index > 30kg/m2
* Arm circumference > 32 cm
* Any condition that may be likely to compromise patients participation to the trial (alcohol or drug abuse, disability illness, etc.)
* Concomitant therapy with antihypertensive drugs non permitted by protocol, corticosteroids or drugs known to affect blood pressure
* Concomitant use of lithium or cholestyramine or colestipol resins (potential drug interactions with HCTZ)
* Investigational drug treatment within the past 30 days before the enrolment or concurrent participation to any other trial
* Sensitivity, significant adverse reaction or contraindications to the study drugs (telmisartan, losartan, HCTZ)
* Predictable lack of patient co-operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2000-01; Primary Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure (DBP) during the last 6 hours (ABPM - ambulatory blood pressure measurement) of the 24-hour dosing interval at the end of the monotherapy period of treatment | Baseline and week 12

SECONDARY OUTCOMES:
Change from baseline in DBP during the last 6 hours (ABPM) of the 24-hour dosing interval at the end of the study | Baseline and week 24
Change from baseline in systolic blood pressure (SBP) during the last 6 hours (ABPM) of the 24-hour dosing interval | Baseline, week 12 and 24
Change from baseline in DBP/SBP during the last 2 hours (ABPM) of the 24-hour dosing interval (trough BP) | Baseline, week 12 and 24
Changes from baseline in trough cuff (sphygmomanometer) SBP/DBP | Baseline, week 12 and 24
Changes from baseline in SBP/DBP of 24 hours mean ABPM | Baseline, week 12 and 24
Comparison of SBP/DBP ABPM tracing profile | Week 12 and 24
Smoothness index in comparison with baseline | Baseline, week 12 and 24
Number of responders | Week 12 and 24
Number of controlled responders | Week 12 and 24
Number of patients who withdraw due to lack of efficacy | 24 weeks
Number of patients with adverse events | 24 weeks
Number of patients who withdraw due to adverse events | 24 weeks